CLINICAL TRIAL: NCT00125333
Title: A Phase 1/2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Safety of Repeated Topical Application of Three Concentrations of NF-kappaB Decoy in Adults With Mild-to-Moderate Atopic Dermatitis
Brief Title: Topical NF-kappaB Decoy in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Responsible Party: Shaun Comfort, MD, Anesiva, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110-01P
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis, eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — NF-kappaB decoy

INTERVENTIONS:
Drug: NF-kappaB Decoy

SUMMARY:
The purpose of this study is to determine whether this topical NF-kappaB Decoy candidate is safe in persons with atopic dermatitis. Preliminary evidence of efficacy (whether it is working) will also be evaluated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to evaluate the safety of repeated application of three concentrations of NF-kappaB Decoy in approximately 75 subjects with mild-to-moderate atopic dermatitis. The face, hands, feet, scalp, or groin may NOT be treated.

Other treatment agents are currently available for atopic dermatitis but present significant potential side effects (topical steroids) or are potent immunosuppressives (topical calcineurin inhibitors) with pending longer-term safety data.

NF-kappaB Decoy is a double-stranded deoxyribonucleic acid (DNA) oligodeoxynucleotide that mimics the NF-kappaB binding sequence on the chromosomal DNA, thereby inhibiting the production of the inflammatory response triggered by NF-kappaB. This mechanism of action presents a unique treatment modality.

A comprehensive series of nonclinical data have produced promising results.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 through 65 years of age and sign an informed consent
* Have been given a diagnosis of mild to moderate atopic dermatitis as defined by: *Pruritus; *Eczematous dermatitis (acute, subacute, chronic) involving at least current or prior flexural lesions with chronic or relapsing course; *Early age of onset (prior to 10 years of age, by history); *Personal or family history of atopy
* If receiving antihistamines, are on a stabilized dose, and expect to maintain this dose throughout the study
* Are females or males of reproductive potential who are compliant in using adequate birth control or are females or males not of reproductive potential

Exclusion Criteria:

* Have concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug
* Have immunocompromised status (such as known human immunodeficiency virus infection)
* Have any clinically significant abnormal clinical laboratory test results at Screening
* Have a history of malignancy not in remission for at least 5 years excluding basal cell carcinoma and nonperiorificial squamous cell carcinoma of the skin
* Have an active intercurrent infection
* Have applied any topical medication (including corticosteroid, calcineurin inhibitor, topical H1 and H2 antihistamines, topical antimicrobials, other medicated topical agents) or herbal preparation to the area selected for treatment within 1 week of the Day 1 visit; have used any systemic antibiotic within 1 week prior to the Day 1 visit; have used any systemic treatment for atopic dermatitis (including systemic corticosteroids, nonsteroidal immunosuppressants, or treatment with light) within 4 weeks prior to the Day 1 visit; have used an investigational drug for any reason within 4 weeks of the Day 1 visit; have used intranasal and/or inhaled corticosteroids at doses > 2 mg prednisone or equivalent per day within 4 weeks of the Day 1 visit; or have used immunosuppressive or immunomodulating drugs such as etanercept, alefacept, or infliximab within 16 weeks prior to Day 1
* Have a history of hypersensitivity or allergic reactions to parabens or any other ingredient in the vehicle formulation
* If female, are pregnant or lactating, or intend to become pregnant during the study period
* If male, have a female partner who is pregnant or lactating, or intends to become pregnant during the study period
* Have any reason which, in the opinion of the investigator, interferes with the ability of the subject to participate in or complete the trial, or which places the subject at undue risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of twice-daily topical application of three concentrations of NF-kappaB Decoy in adult subjects with mild-to-moderate atopic dermatitis

SECONDARY OUTCOMES:
To make a preliminary evaluation of the efficacy of the topical NF-kappaB Decoy in the treatment of mild-to-moderate atopic dermatitis in adult subjects
To evaluate the systemic pharmacokinetic (PK) profile of NF-kappaB Decoy

CONTACTS AND LOCATIONS:
Overall Officials: Andria Langenberg, MD, Study Director — Anesiva, Inc.
Locations (9):
- United States (9):
  - University of Miami Skin Research, Miami, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Helendale Dermatology & Medical Spa, LLP, Rochester, New York
  - Oregon Health & Science University, Department of Dermatology, Portland, Oregon
  - Derm Research, Inc., Austin, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, South Houston, Texas
  - Madison Skin & Research, Inc., Madison, Wisconsin